CLINICAL TRIAL: NCT06541691
Title: Coated or Chewable Aspirin in Patients with Established Atherosclerotic Disease and a Hybrid Strategy to Mitigate the Adverse Effects of Air Pollution: the COATED-AIR Randomized Clinical Trial
Brief Title: Coated or Chewable Aspirin and a Hybrid Strategy to Mitigate Adverse Effects of Air Pollution in Stable Atherosclerotic Disease
Acronym: COATED-AIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Parham Sadeghipour, Dr., Rajaie Cardiovascular Medical and Research Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4020310
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-08

CONDITIONS: Atherosclerotic Cardiovascular Disease; Coronary Artery Disease; Ischemic Heart Disease; Ischemic Stroke; Peripheral Arterial Disease; Carotid Artery Stenosis; Carotid Atherosclerosis
Keywords: atherosclerosis; atherosclerotic cardiovascular disease; atherosclerotic arterial disease; atherosclerotic plaque; coronay artery disease; ischemic heart disease; atherosclerotic disease; ischemic stroke; peripheral arterial disease; carotid artery stenosis; carotid atherosclerosis; myocardial infarction; acute limb ischemia; bleeding; major bleeding; gastrointestinal bleeding; gastrointestinal ulcer; peptic ulcer disease; gastric ulcer; duodenal ulcer; dyspepsia; intracerebral hemorrhage; aspirin; acetylsalicylic acid; antithrombotic therapy; antithrombotic agents; antiplatelet agents; air pollution; cerebral hemorrhage; hemorrhage
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Myocardial Ischemia; Ischemic Stroke; Peripheral Arterial Disease; Carotid Stenosis; Carotid Artery Diseases; Plaque, Atherosclerotic; Myocardial Infarction; Hemorrhage; Gastrointestinal Hemorrhage; Peptic Ulcer; Stomach Ulcer; Duodenal Ulcer; Dyspepsia; Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: 2×2 full factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The quadruple masking (Participant, Treating Clinician, Investigator, Outcomes Assessor) is used for the first randomization, and the second randomization is open-label with blinded adjudication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Enteric-coated aspirin (+/- hybrid strategy) (Experimental): 81 mg enteric-coated aspirin (+/- a hybrid strategy to mitigate the cardiovascular adverse effects of the air pollution)
  Interventions: Drug: Enteric-coated aspirin
- Plain aspirin (+/- hybrid strategy) (Active Comparator): 81 mg plain aspirin (+/- a hybrid strategy to mitigate the cardiovascular adverse effects of the air pollution)
  Interventions: Drug: Plain aspirin
- Hybrid strategy (with enteric-coated or plain aspirin) (Experimental): A hybrid strategy to mitigate the cardiovascular adverse effects the air pollution, composed of one-page educational flashcard, cell phone text messages alerting participants on polluted days, recommending them to stay indoors or wear KN-95 facemasks provided by the study team in case of necessary outdoor activity, and recommendation to consume citrus fruits on polluted days.
  Interventions: Other: Hybrid strategy
- Usual care (with enteric-coated or plain aspirin) (No Intervention): No active strategy (usual care) without any clear recommendations related to air pollution; only a control card will be shared with the patients randomized to the usual care

INTERVENTIONS:
Drug: Enteric-coated aspirin — Enteric-coated aspirin tablet 81 mg, once daily
  Other Names: Low dose of enteric-coated aspirin
  Arms: Enteric-coated aspirin (+/- hybrid strategy)
Drug: Plain aspirin — Plain aspirin tablet 81 mg, once daily
  Other Names: Low dose of plain aspirin
  Arms: Plain aspirin (+/- hybrid strategy)
Other: Hybrid strategy — A hybrid strategy composed from:
  * A one-page educational flashcard
  * Alerting patients on highly polluted days via text message
  * Encouraging patients to stay at home or minimizing outdoor activity on highly polluted days
  * Encouraging patients via text message to wear KN-95 facemasks (provided by the investigators of this study) during outdoors time on highly polluted days
  * Encouraging patients to consume citrus fruits during highly polluted days
  Other Names: The hybrid strategy to mitigated the cardiovascular adverse effects of the air pollution
  Arms: Hybrid strategy (with enteric-coated or plain aspirin)

SUMMARY:
Although both enteric-coated and plain formulations of aspirin are being used commonly, there are no high-quality comparisons between these formulations with respect to clinical efficacy outcomes in patients with atherosclerotic cardiovascular diseases (ASCVD). Air pollution is also a major contributor to the excess risk of cardiovascular events in many regions of the world. However, little is known about the effect of individual-level mitigation strategies against air pollution in reducing cardiovascular outcomes. The purpose of the first randomization is to compare the efficacy and safety of enteric-coated versus plain low-dose (81 mg) aspirin formulations in a double-blind fashion. The second randomization compares a multifaceted intervention including one-page educational flashcard, cell phone text messages alerting participants on polluted days, recommending them to stay indoors or wear KN-95 facemasks provided by the study team in case of necessary outdoor activity, and recommendation to consume citrus fruits on polluted days versus usual care. Both randomization are powered for clinical outcomes and the results will inform practice.

DETAILED DESCRIPTION:
- Background: Aspirin is a key treatment option of patients with atherosclerotic cardiovascular disease (ASCVD). The enteric coating has emerged as a potential solution to minimize the exposure of the gastric mucosa to the medication. However, change in the medication main site of absorption might negatively impact the pharmacokinetics/pharmacodynamics of aspirin and alter its antithrombotic properties, leading to diminished efficacy of the medication. A sufficiently large randomized controlled trial with a long-term follow-up to compare the effectiveness of enteric-coated versus plain aspirin in reducing adverse cardiovascular events and mitigating the adverse effects of the medication in patients with ASCVD is lacking.

Ambient air pollution is a prominent cause of mortality, being associated with 6.7 million deaths worldwide every year, half of which are attributable to cardiovascular causes. Near the half of these deaths is attributable to cardiovascular causes. Several patient-level interventions have been proposed to counteract with the adverse effects of the air pollution, including alerting patients via text message, staying at home, using face masks, or consuming citrus fruits (as a source of vitamin C) during the days with air pollution. However, the effect of implementing these strategies, individually and especially as a group, in mitigating the adverse effects of the air pollution has not yet been studied in a randomized controlled trial powered for clinical outcomes.

The purpose of the current randomized clinical trial is to compare the efficacy and safety of enteric-coated versus plain low-dose (81 mg) aspirin formulations in a double-blind fashion, and an open-label comparison of a multifaceted intervention including a one-page informational flashcard, cell phone message alerting on days with poor air quality to encourage patients not to spend time outdoors or to wear KN-95 facemasks outdoors in those days, and encouraging patients to consume citrus fruits on highly polluted days (hereafter referred to as hybrid strategy), versus usual care, in a multicenter randomized controlled trial (RCT) with a 2x2 factorial design.

- Design and Randomization method: Multicenter randomized controlled trial with a 2x2 full factorial design with double-blind randomization with a 1:1 allocation ratio to low-dose enteric-coated vs plain aspirin, and open-label randomization with 1:1 allocation ratio to hybrid strategy to reduce the cardiovascular effects of air pollution vs usual care. Permuted block randomization with block sizes of 8, 12 and 16 chosen randomly via an electronic web-based system will be used for the study. The allocation sequence will be concealed. All outcomes will be adjudicated by a Clinical Events Committee blinded to the assigned treatments.

- Setting: Teaching hospitals in Tehran province, Iran will be involved.

- Statistical consideration and sample size calculation: An event-driven approach was considered for the calculation of sample size. Considering a relative hazard reduction of 23% in the first (aspirin formulation) randomization and 25% in the second (air pollution mitigation strategy) randomization, to provide a two-sided alpha of 0.05 and a statistical power of 80%, a total number of 460 primary efficacy outcomes for the first randomization and 380 primary efficacy outcomes for the second randomization would be needed. An event-rate of 18.5% for the incidence of primary efficacy outcome in the control arm of the first randomization, and 19.2% for the incidence of primary efficacy outcome in the control arm of the second randomization was assumed per a median follow-up of 2-year. Ultimately, Considering 4% dropout rate per each randomization, a total number of 2920 and 2732 patients would be needed for the first and second randomizations, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with documented ASCVD defined as at least one of the following:

  * Coronary artery disease (CAD):

    1. Previous or recent documented type I myocardial infarction *(if not specified, will be assumed as type I)
    2. History of coronary revascularization (percutaneous coronary intervention or coronary artery bypass graft surgery)
    3. History of obstructive CAD (>50% stenosis) documented by coronary computed tomography (CT) or conventional angiography
  * Peripheral arterial disease (PAD):

    1. Previous or recent acute ischemic limb event (>7 days prior)
    2. History of previous endovascular/surgical lower or upper extremities revascularization for an atherosclerotic cause
    3. History of ulcer or lower extremities amputation due to ASCVD.
  * Carotid arterial diseases:

    1. History of previous endovascular/surgical carotid artery revascularization for atherosclerotic causes
    2. History of > 50% carotid artery stenosis based on documented imaging tests (Duplex US, CT angiography, magnetic resonance angiography, or conventional angiography)
  * Ischemic stroke:

    1. History of recent or previous documented ischemic stroke not due to atrial fibrillation, endocarditis, or systemic hypoperfusion/hypotension, being treated with low-dose aspirin
* Inhabitant of Tehran province
* Willing to participate and able to provide written informed consent

Exclusion Criteria:

* Being within 72 days of acute/unstable atherosclerotic cardiovascular events (acute myocardial infarction, acute limb event, and acute ischemic stroke), or within 72 hours of revascularization.
* Patients receiving triple antithrombotic therapy
* History of upper gastrointestinal bleeding within the past 30 days
* History of intracranial hemorrhage within the past 30 days
* End-stage kidney disease with estimated creatinine clearance < 15 mL/min, or undergoing hemodialysis or peritoneal dialysis
* Known comorbidities associated with poor prognosis (e.g., metastatic cancer) in conjunction with an estimated life expectancy of less than one year according to the treating clinician
* Any other conditions that make the participants unsuitable for recruitment or follow-up (e.g., illiteracy)
* Not having aspirin as part of the planned durable treatment regimen
* Inability to receive/read text messages/phone calls by personal mobile phone (or that of a caregiver who lives with the patient and is willing to relay messages)

  * The full list of exclusion criteria is provided in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Composite of fatal or nonfatal ischemic stroke (not deemed to be related to systemic hypotension), type I myocardial infarction, and acute limb events | within maximum of 30-month follow-up
  Time to the first occurrence of an outcome composed of any endpoint that fulfills the definite criteria for diagnosis of at least one of the ischemic stroke, type I myocardial infarction, or acute limb event (whether leading to the patient's death or not) as defined in the description of the related secondary outcomes This outcome is assigned as the primary efficacy outcome for the first randomization.
Composite of non-fatal ischemic stroke (not deemed to be related to systolic hypotension), type I myocardial infarction, acute limb events, or cardiovascular death | within maximum of 30-month follow-up
  Time to the first occurrence of an outcome composed of any endpoint that fulfills the definite criteria for diagnosis of at least one of the ischemic stroke, type I myocardial infarction, or acute limb event, and don not result in patient death as defined in the description of the related secondary outcomes This outcome is assigned as the primary outcome for the second randomization.

SECONDARY OUTCOMES:
Type I myocardial infarction | within maximum of 30-month follow-up
  Time to the first occurrence of type I myocardial infarction. Type I myocardial infarction is defined as spontaneous clinical syndrome related to atherosclerotic plaque rupture, ulceration, fissuring, erosion, or dissection, with resulting intraluminal thrombus and leading to decreased myocardial blood flow or distal platelet emboli with ensuing myocyte necrosis. This classification requires the detection of a rise and/or fall of cardiac biomarker values (preferably cTn) with at least 1 value >99th percentile of the URL and at least 1 of the following: 1- Symptoms of myocardial ischemia 2- New or presumed new significant ST-segment T wave changes or new left bundle branch block on the ECG 3- Development of pathological Q waves on the ECG 4- Imaging evidence of new loss of myocardium or new regional wall motion abnormality 5- Identification of an intracoronary thrombus by angiography or autopsy
Ischemic stroke (not deemed to be related to systemic hypotension) | within maximum of 30-month follow-up
  Time to the first occurrence of ischemic stroke. Ischemic stroke is defined as an episode of acute neurological dysfunction caused by focal cerebral, spinal, or retinal infarction as a result of arterial thrombosis and/or thromboembolism (not deemed to be related to systemic hypotension/hypoperfusion), and lasting ≥ 24 hours or to time of death with residual neurological sequelae
Acute limb event | within maximum of 30-month follow-up
  A limb-threatening ischemia that is confirmed by limb hemodynamics or imaging and leads to an acute vascular intervention (i.e., pharmacologic [heparin, thrombolysis], peripheral arterial surgery/reconstruction, peripheral angioplasty/stenting, and/or limb amputation) within 30 days of onset of symptoms. In case of lack of confirmation by limb hemodynamics or imaging, the absence of pedal pulses is acceptable as the hemodynamic criterion for acute limb ischemia
All-cause death | within maximum of 30-month follow-up
  Death due to any causes (cardiovascular, non-cardiovascular, or undetermined) within the follow-up period
Cardiovascular death | within maximum of 30-month follow-up
  Cardiovascular death is defined as death resulting from cardiovascular causes. The following categories may be collected: 1- Death caused by acute MI 2- Death caused by sudden cardiac, including unwitnessed, death 3- Death resulting from heart failure 4- Death caused by stroke 5- Death resulting from cerebrovascular hemorrhage 6- Death resulting from other cardiovascular causes such as PE, acute aortic syndromes, arrhythmia, and others
Unplanned vascular hospitalization | within maximum of 30-month follow-up
  Inpatient admission to a hospital specifically due to acute events involving the vascular system. This encompasses conditions such as acute myocardial infarction, ischemic or hemorrhagic stroke, acute limb ischemia, and other vascular emergencies necessitating urgent medical care and hospitalization
Composite of International Society on Thrombosis and Haemostasis (ISTH) major or clinically-relevant non-major gastrointestinal (GI) bleeding that bleeding and new symptomatic diagnosed gastroduodenal ulcer | within maximum of 30-month follow-up
  Time to the first occurrence of an outcome composed of any GI bleeding that fulfills the ISTH criteria for major or clinically-relevant non-major bleeding (defined in the description of the related secondary outcomes), and/or any newly diagnosed symptomatic gastroduodenal ulcer that meets the definition described in the description of the related secondary outcomes.
  This outcome is considered as the primary safety outcome for the first randomization.
Upper GI bleeding | within maximum of 30-month follow-up
  Bleeding originating from sites in the esophagus, stomach, or duodenum with manifestations including hematemesis (vomiting of red blood or coffee-grounds material), melena (black, tarry stool), or hematochezia (passage of red or maroon material per rectum). Major and clinically relevant non-major UGIB will also be discriminated.
Clinically relevant non-major GI bleeding | within maximum of 30-month follow-up
  Bleeding from the upper or lower gastrointestinal tract that meets the criteria for the ISTH definition for clinically-relevant non-major bleeding (Please see below for these two definitions).
Any Major bleeding | within maximum of 30-month follow-up
  Any bleeding event fulfills the ISTH major bleeding criteria in non-surgical patients defined as having a symptomatic presentation and: 1- Fatal bleeding and/or 2- Bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome and/or 3- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Intracranial hemorrhage | within maximum of 30-month follow-up
  The abnormal bleeding within the confines of the skull, involving either the brain tissue (intracerebral hemorrhage) or the spaces between the layers that cover the brain (subarachnoid or subdural hemorrhage).
Any clinically relevant non-major bleeding | within maximum of 30-month follow-up
  Any sign or symptom of hemorrhage (e.g., more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria: 1- Requiring medical intervention by a healthcare professional 2- Leading to hospitalization or increased level of care 3- Prompting a face-to-face (i.e., not just a telephone or electronic communication) evaluation.
New symptomatic diagnosed gastroduodenal ulcer | within maximum of 30-month follow-up
  Gastroduodenal ulcer manifested by gastrointestinal symptoms that persist for > 3 days, with confirmation of ulcer by endoscopy. An ulcer is defined as any mucosal break at least 3 mm in greatest diameter

CONTACTS AND LOCATIONS:
Overall Officials: Parham Sadeghipour, M.D, Principal Investigator — Rajaie Cardiovascular Medical and Research Center
Locations (1):
- Rajaie Cardiovascular Medical and Research Center, Tehran, Tehran Province, Iran